CLINICAL TRIAL: NCT03318224
Title: Fatigue in Germany - Examination of Prevalence, Severity, and State of Screening and Treatment
Brief Title: Fatigue Prevalence, Severity, and State of Treatment in Germany
Acronym: FiX
Status: Completed | Type: Observational
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: FiX
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cancer-related Fatigue
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: none (observational study) — only assessments via questionnaires, no interventions

SUMMARY:
Fatigue is a major concern during and after cancer therapy with severe impact on quality of life. Yet, sound comparable data on fatigue prevalence, severity, and impact on daily life across different tumor entities is lacking. Furthermore, little is known about the current state of screening, counselling and treatment of fatigue.

Thus, the FiX-Study aims to assess such data to identify patient groups with especial need for an improved fatigue management and treatment.

A minimum of n=3000 patients about equally distributed about the 16 most common tumor entities shall be recruited between year 1 and 2 after primary cancer diagnosis via the cancer registry Baden-Württemberg. Data on fatigue (EORTC QLQ-FA12, BFI), quality of life (EORTC QLQ-C30), depression and anxiety (PAQ-4), and information about screening and treatment of fatigue will be assessed via self-reported questionnaires. Clinical data regarding tumor and treatment characteristics will be derived from the cancer registry.

This trial is imbedded in a larger research agenda on fatigue and will provide the basis for the development of an individually-tailored fatigue program.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of Age
* Diagnosed with a primary tumor of one of the following malignant neoplasms (including in-situ carcinoma): stomach (C16, D00.2), colon (C18, D01.0), rectum (C19-20, D01.1-1.2), liver (C22, D01.5), pancreas (C25, D01.7), lung (C33-34, D02.1-2.2), malignant melanoma (C43, D03), breast (C50, D05, female only), cervix or ovaries (C53, D06), endometrium (C54.1, D07.0), ovaries (C56), prostate (C61), kidney (C64), bladder (C67, D09.0), non-Hodgkin lymphoma (C82-88), leukemia (C91-C95)
* Time since first diagnosis is at least 1 year, maximal 2 years
* Able to understand and follow the study protocol.

Exclusion Criteria:

• Any additional malignant or unclear neoplasm or carcinoma in situ at or since time of diagnosis of the considered primary tumor, except non-malignant, unspecified, or in-situ neoplasm of skin (C44 or D0.4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who were diagnosed 1-2 years ago
Sampling Method: Probability Sample
Enrollment: 2508 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
EORTC QLQ-FA12 | Assessment time point: about 1-2 years post-diagnosis
  12-item multidimensional fatigue questionnaire
Brief Fatigue Inventory (BFI) | Assessment time point: about 1-2 years post-diagnosis
  Questionnaire on the impact of fatigue

SECONDARY OUTCOMES:
EORTC QLQ-C30 | Assessment time point: about 1-2 years post-diagnosis
  Quality of Life questionnaire
PHQ-4 | Assessment time point: about 1-2 years post-diagnosis
  Anxiety and Depression Screen
State of fatigue management | Assessment time point: about 1-2 years post-diagnosis
  Questionnaire on Screening, primary evaluation, and received counseling, treatment and interventions for fatigue
Patient's believes and knowledge with regard to fatigue | Assessment time point: about 1-2 years post-diagnosis
  7 Likert-items regarding believes and knowledge about fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- German Cancer Research Center, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schmidt ME, Hermann S, Arndt V, Steindorf K. Prevalence and severity of long-term physical, emotional, and cognitive fatigue across 15 different cancer entities. Cancer Med. 2020 Nov;9(21):8053-8061. doi: 10.1002/cam4.3413. Epub 2020 Sep 7. PMID 32893501
- [Background] Schmidt ME, Bergbold S, Hermann S, Steindorf K. Knowledge, perceptions, and management of cancer-related fatigue: the patients' perspective. Support Care Cancer. 2021 Apr;29(4):2063-2071. doi: 10.1007/s00520-020-05686-5. Epub 2020 Aug 29. PMID 32860177
- [Derived] Schmidt ME, Blickle P, Steindorf K. Cancer-related fatigue: Identification of hallmarks to enable refined treatment approaches. Psychooncology. 2022 Dec;31(12):2169-2176. doi: 10.1002/pon.6061. Epub 2022 Nov 9. PMID 36314131